CLINICAL TRIAL: NCT01980927
Title: Changes in Intracranial Compliance in Migraine Subjects Following a National Upper Cervical Chiropractic Association (NUCCA)Atlas Correction Intervention - a Pilot Study
Brief Title: Changes in Intracranial Compliance in Migraine Subjects Following a National Upper Cervical Chiropractic Association Atlas Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Werner Becker, Dr. Werner Becker, MD, FRCPC, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24116
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Migraine
Keywords: Migraine; National Upper Cervical Chiropractic Association atlas correction
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NUCCA atlas correction (Experimental): NUCCA atlas correction for migraine patients
  Interventions: Procedure: NUCCA atlas correction

INTERVENTIONS:
Procedure: NUCCA atlas correction — A chiropractic procedure involving correcting a misalignment of the atlas or "top" vertebra in the spine.

SUMMARY:
A small number of chiropractors, who align only the atlas C-1, or "top" vertebra in the spine, practice the National Upper Cervical Chiropractic Association (NUCCA) atlas correction procedure. This procedure uses a precise, non-invasive, gentle touch technique to correct misalignment of the atlas. Although NUCCA practitioners have long used this procedure in the treatment of headache, it has not been formally studied using clinical trials. There is some data indicating that NUCCA correction can increase intracranial compliance. This intracranial compliance can be measured by a magnetic resonance imaging (MRI) study before and then after a NUCCA procedure. In this study, the investigators hope to show that the correction of an atlas misalignment will increase intracranial compliance in subjects with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-65 years of age.
* Be naive to Upper Cervical Chiropractic care. Other forms of chiropractic care in the past are permitted.
* Have migraine with or without aura.
* Have between 10-26 headache days per month over the last 4 months.
* Have at least 4 separate headache episodes per month, with episodes separated by at least 4 hours of painfree time.
* Have at least 8 days per month with pain of levels greater than or equal to 4/10 for part of the day, or have attacks successfully treated with migraine specific medication.
* Be candidates suitable for NUCCA therapeutic intervention because of atlas displacement as assessed by NUCCA investigator.
* Subjects on acceptable pharmacological prophylaxis must either remain on a stable dose throughout the study, or stop the prophylactic medication one month before entering the baseline period.

Exclusion Criteria:

* Any medical or psychiatric condition which in the opinion of the investigator would make the subject unsuitable for enrolment, because of inability to comply with study requirements or possible confounding of the results.
* Headache on more than 26 days per month.
* Acute medication overuse as defined by the International Classification of Headache Disorders.
* Pregnancy or lactation
* Severe cervical spine degeneration as assessed by cervical spine x-ray.
* Claustrophobia or any condition that contraindicates an MRI scan
* A history of cardiovascular disease, cerebrovascular disease, brain surgery, or other central nervous system disorder.
* Other chronic pain disorder which might interfere with headache assessment or study procedures.
* A history of significant hypo- or hypertension as determined by the investigator.
* Subject on a beta-blocker, calcium channel blocker, or other medication which the investigator considers might alter cerebral vascular regulation. Triptans are allowed, but must not be taken within 24 hours (48 hours for frovatriptan) before an MRI study.
* A history of substance abuse or dependence within 1 year.
* Current participation in a research study or within the last 30 days.
* Any spinal chiropractic care outside of the study protocol is prohibited during the baseline and treatment period.
* Use of botulinum A within 4 months of study entry.
* A history of significant head or neck trauma (as judged by the investigator) within the year prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in intracranial compliance; comparing the baseline period to one month post treatment, 4 weeks after initiation of NUCCA care and maintained correction of atlas misalignment, as measured by phase contrast magnetic resonance imaging. | At baseline, at 4 weeks, at 8 weeks

SECONDARY OUTCOMES:
Days with headache per month | At baseline, at 4 weeks, at 8 weeks
  Patients use headache diaries to track the number of days with headaches.
Average headache intensity on headache days | At baseline, at 4 weeks, at 8 weeks
  Patients rate headache pain from 0-10 on 3 segments of the day (morning, afternoon, evening) using headache diaries. These numbers are used to calculate the average intensity of the headache on headache days.

OTHER OUTCOMES:
Quality of life measurements - comparing quality of life scores by using various questionnaires at baseline and at 8 weeks | At baseline, at 8 weeks
  Using MIDAS, Migraine QOL, and HIT-6 questionnaires to score patients' quality of life in measurable terms.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Becker, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Woodfield HC 3rd, Hasick DG, Becker WJ, Rose MS, Scott JN. Effect of Atlas Vertebrae Realignment in Subjects with Migraine: An Observational Pilot Study. Biomed Res Int. 2015;2015:630472. doi: 10.1155/2015/630472. Epub 2015 Dec 10. PMID 26783523